CLINICAL TRIAL: NCT01596673
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Assess the Abuse Potential of the Hydrocodone Bitartrate Extended-Release Tablet in Healthy, Nondependent, Recreational Opioid Users
Brief Title: A Study to Assess the Abuse Potential of Hydrocodone Extended-Release Tablet in Recreational Opioid Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C33237/1085
Record Dates: First submitted 2012-03-30; First posted 2012-05-11 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Hydrocodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BCAD Treatment Group (Experimental): Subjects in this group will receive study drug in the following sequence:
  Treatment B - 1 intact placebo tablet, hydrocodone bitartrate powder at a dose strength of 45 mg reconstituted in 60 mL of a noncarbonated flavored beverage, and 1 crushed placebo tablet.
  Treatment C - 1 intact 45-mg hydrocodone bitartrate extended-release tablet, 60 mL of a noncarbonated flavored beverage, and 1 crushed placebo tablet.
  Treatment A - 1 intact placebo tablet, 60 mL of a noncarbonated flavored beverage, 1 crushed 45-mg hydrocodone bitartrate extended-release tablet.
  Treatment D - 1 intact placebo tablet, 60 mL of a noncarbonated flavored beverage, and 1 crushed placebo tablet(matching the 45-mg hydrocodone bitartrate extended-release tablet).
  Interventions: Drug: 45-mg hydrocodone bitartrate extended-release tablet (crushed or intact); Drug: Placebo
- CDBA Treatment Group (Experimental): Subjects in this group will receive study drug in the following sequence:
  Treatment C - 1 intact 45-mg hydrocodone bitartrate extended-release tablet, 60 mL of a noncarbonated flavored beverage, and 1 crushed placebo tablet.
  Treatment D - 1 intact placebo tablet, 60 mL of a noncarbonated flavored beverage, and 1 crushed placebo tablet (matching the 45-mg hydrocodone bitartrate extended-release tablet).
  Treatment B - 1 intact placebo tablet, hydrocodone bitartrate powder at a dose strength of 45 mg reconstituted in 60 mL of a noncarbonated flavored beverage, and 1 crushed placebo tablet.
  Treatment A - 1 intact placebo tablet, 60 mL of a noncarbonated flavored beverage, 1 crushed 45-mg hydrocodone bitartrate extended-release tablet.
  Interventions: Drug: 45-mg hydrocodone bitartrate extended-release tablet (crushed or intact); Drug: Placebo
- DACB Treatment Group (Experimental): Subjects in this group will receive study drug in the following sequence:
  Treatment D - 1 intact placebo tablet, 60 mL of a noncarbonated flavored beverage, and 1 crushed placebo tablet(matching the 45-mg hydrocodone bitartrate extended-release tablet).
  Treatment A - 1 intact placebo tablet, 60 mL of a noncarbonated flavored beverage, 1 crushed 45-mg hydrocodone bitartrate extended-release tablet.
  Treatment C - 1 intact 45-mg hydrocodone bitartrate extended-release tablet, 60 mL of a noncarbonated flavored beverage, and 1 crushed placebo tablet.
  Treatment B - 1 intact placebo tablet, hydrocodone bitartrate powder at a dose strength of 45 mg reconstituted in 60 mL of a noncarbonated flavored beverage, and 1 crushed placebo tablet.
  Interventions: Drug: 45-mg hydrocodone bitartrate extended-release tablet (crushed or intact); Drug: Placebo
- ABDC Treatment Group (Experimental): Subjects in this group will receive study drug in the following sequence:
  Treatment A - 1 intact placebo tablet, 60 mL of a noncarbonated flavored beverage, 1 crushed 45-mg hydrocodone bitartrate extended-release tablet.
  Treatment B - 1 intact placebo tablet, hydrocodone bitartrate powder at a dose strength of 45 mg reconstituted in 60 mL of a noncarbonated flavored beverage, and 1 crushed placebo tablet.
  Treatment D - 1 intact placebo tablet, 60 mL of a noncarbonated flavored beverage, and 1 crushed placebo tablet(matching the 45-mg hydrocodone bitartrate extended-release tablet).
  Treatment C - 1 intact 45-mg hydrocodone bitartrate extended-release tablet, 60 mL of a noncarbonated flavored beverage, and 1 crushed placebo tablet.
  Interventions: Drug: 45-mg hydrocodone bitartrate extended-release tablet (crushed or intact); Drug: Placebo

INTERVENTIONS:
Drug: 45-mg hydrocodone bitartrate extended-release tablet (crushed or intact) — Phase B:
  Eligible subjects will be randomized to treatment sequence XY or YX whereby treatment X is 60 mL of a noncarbonated flavored beverage and treatment Y is hydrocodone bitartrate powder at a dose strength of 45-mg reconstituted in 60 mL of a noncarbonated flavored beverage.
  Phase C:
  Eligible subjects will be randomly assigned to 1 of 4 treatment arms:
  Treatment A: intact placebo tablet, 60 mL noncarbonated flavored beverage, 1 crushed 45-mg hydrocodone bitartrate extended-release tablet.
  Treatment B: intact placebo tablet, hydrocodone bitartrate powder at a dose strength of 45-mg in 60 mL of a noncarbonated flavored beverage and 1 crushed placebo tablet.
  Treatment C: intact 45-mg hydrocodone bitartrate extended-release tablet, 60 mL noncarbonated flavored beverage, and 1 crushed placebo tablet Treatment D: intact placebo tablet, 60 mL noncarbonated flavored beverage, and 1 crushed placebo tablet.
  Other Names: hydrocodone
Drug: Placebo — Placebo will consist of 60 mL of a non-carbonated beverage without the addition of active treatment

SUMMARY:
The purpose of this study is to assess the relative abuse potential of the hydrocodone bitartrate extended-release tablet compared to immediate-release hydrocodone bitartrate.

DETAILED DESCRIPTION:
Hydrocodone bitartrate is a semisynthetic opioid analgesic and antitussive. Hydrocodone is widely used for various indications similar to those of codeine, primarily for relief of moderate to moderately severe pain. For the treatment of pain in the United States, hydrocodone is currently available only as an immediate-release (IR) product in combination with other medications such as acetaminophen or ibuprofen. The extended-release (ER) formulation tested in this study is designed to be resistant to dose dumping with alcohol or rapid release of hydrocodone after tampering.

The study will consist of 3 phases: A, B,and C. Phase A is the screening phase where subject eligibility will be confirmed (Visit 1). Subjects who are eligible will enter Phase B, a double-blind, 2-period crossover design (Visit 2) followed by Phase C, a double-blind 4-period crossover design (Visits 3 through 6).

Phase B is the randomized, double-blind, placebo-controlled, 2-treatment, 2- period crossover portion of the study which is designed to ensure that the subject can tolerate a 45-mg dose of hydrocodone and that the subject can discriminate between the effect of hydrocodone and the effect of placebo. Subjects will arrive at the study center on the day prior to the first study drug administration and remain at the study center for a minimum of 24 hours after the second study drug administration in phase B. After a review of the inclusion/exclusion criteria and check-in procedures (including a Naloxone Challenge),eligible subjects will be randomly assigned to one of 2 treatment sequences. For subjects who qualify to continue into phase C, there will be a minimum 7-day washout period between the second dose in phase B and the first dose in phase C.

Phase C is the randomized, double-blind, triple-dummy, placebo-controlled, 4-period crossover portion of the study. Subjects will arrive at the study center the day prior to each study drug administration in phase C and remain at the study center through 72 hours after study drug administration in each period. Eligible subjects will be randomly assigned to 1 of 4 treatment groups. Each dose in phase C will be separated by a minimum 14 day washout period.

All subjects (including those who withdraw from the study) will be asked to return to the study center for a follow-up visit approximately 48 to 72 hours after discharge from the study center following their final dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained.
* The subject speaks and writes in English.
* The subject is not physically dependent on opioids as demonstrated by successful completion of a naloxone challenge; ie, subject does not exhibit signs or symptoms of opioid withdrawal (as assessed by a Clinical Opiate Withdrawal Scale score of <5) following administration of intravenous naloxone in the Naloxone Challenge.
* The subject has a history of recreational opioid use to achieve a "high" at least 10 times in the last year and at least on 1 occasion within the 12 weeks before screening. Subjects who abuse multiple drugs should express a preference for opioids.
* The subject is aged 18 through 50 years with a minimum body weight of 50 kg and a body mass index (BMI) of 18.0 through 32.0 kg/m2.
* The subject is in good health as determined by medical and psychiatric history, physical examination, ECG, serum chemistry, hematology, urinalysis, and serology.
* The subject, if a woman, is surgically sterile or 2 years postmenopausal, or if of childbearing potential, is currently using a medically accepted method of contraception and agrees to continue use of this method for the duration of the study (and for 30 days after participation in the study). Acceptable methods of contraception include abstinence, or an intrauterine device (known to have a failure rate of less than 1% per year).
* The subject must have a negative urine drug screen (except for tetrahydrocannabinol) and a negative alcohol test at screening. NOTE: If a subject tests negative for tetrahydrocannabinol at screening, the test result at baseline must be negative for the subject to be considered for enrollment in the study.
* The subject is willing to comply with study restrictions and remain at the study center for the duration of each treatment period during the study.

Exclusion Criteria:

* The subject has any clinically significant uncontrolled medical conditions (treated or untreated).
* The subject has a clinically significant deviation from normal in the clinical laboratory values or ECG or physical examination findings, as determined by the investigator or the medical monitor.
* The subject is a poor metabolizer of cytochrome P450 (CYP2D6) substrates based on genotyping performed at screening.
* The subject currently or has habitually consumed, within the past 2 years, more than 28 units of alcohol per week for male subjects or 21 units of alcohol per week for female subjects, or has a history or current diagnosis of substance dependence as assessed using by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR). NOTE: A unit of alcohol is equal to 1 ounce of hard liquor, 5 ounces of wine, or 8 ounces of beer.
* The subject has participated in, is currently participating in or is seeking treatment for substance-related disorders (excluding nicotine).
* The subject is a heavy smoker (>20 cigarettes per day), chews tobacco and/or is unable to abstain from smoking for 6 hours during any day, or abstain from caffeine intake for 20 hours during any day.
* The subject is a pregnant or lactating woman. (Any woman becoming pregnant during the study will be withdrawn from the study.)
* The subject has previously participated in a Cephalon-sponsored clinical study with the hydrocodone bitartrate extended-release tablet.
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery [appendectomy allowed]).
* The subject has a known sensitivity or idiosyncratic reaction to any compound present in hydrocodone or hydromorphone, their related compounds, or to any metabolites, to the solution used for reconstitution of the immediate-release product, or to any compound listed as being present in a study formulation or naloxone.
* The subject has received any investigational drug within 30 days or 5 half-lives (whichever is longer) before the first study drug administration in phase B.
* The subject has used any vitamins within 2 weeks before the first study drug administration in phase B or has used any systemic or topical prescription, or nonprescription medication (ie, over-the-counter [OTC] medications [except acetaminophen or ibuprofen]) within 2 weeks before the first study drug administration in phase B without evaluation and approval from the medical monitor.
* The subject has used herbal supplements within 2 weeks before the first study drug administration in phase B without evaluation and approval from the medical monitor.
* The subject has donated any plasma within 7 days prior to screening.
* The subject has donated any blood in excess of 450 mL within 56 days prior to screening.
* The subject has, after resting for 5 minutes, elevated blood pressure (defined as seated systolic blood pressure of equal to or more than 140 mm Hg and/or seated diastolic blood pressure of equal to or more than 90 mm Hg), or has hypotension (defined as seated systolic blood pressure of less than 90 mm Hg and/or seated diastolic blood pressure of less than 45 mm Hg). NOTE: No more than 2 rechecks of the subject's blood pressure are permitted at screening.
* The subject has, after resting for 5 minutes, a seated pulse outside the range of 45 to 90 bpm. NOTE: No more than 2 rechecks of the subject's pulse are permitted at screening.
* The subject has, after resting for 5 minutes, oxygen saturation less than 95%. NOTE: No more than 2 rechecks of the subject's SpO2 are permitted for eligibility purposes.
* The subject has a recent history of disclosed violence and/or disclosure of probation/parole.
* The subject has, within 2 weeks before the first dose of study drug in phase B, a clinically significant excessive consumption of coffee, tea, and/or other caffeine-containing beverage or food (ie, 1000 mg of caffeine or more per day, or 8 or more cups of coffee per day).
* The subject has, within 4 weeks before the first study drug administration in phase B, a clinically significant illness or, within 1 week before the first study drug administration in phase B, has any acute illness, or at screening or on the day before the first study drug administration in phase B, has symptoms of any clinically significant or acute illness.
* The subject is unlikely to comply with the study protocol or is unsuitable for any other reason, as judged by the investigator.
* The subject has a positive test result for hepatitis B surface antigen (HBsAg) or antibodies to hepatitis C.
* The subject has a known positive history of antibodies to human immunodeficiency virus (HIV) or HIV disease
* The subject has a clinical laboratory test value(s) outside the following range(s), or any other clinically significant laboratory abnormality as determined by an investigator or medical monitor:
* hemoglobin value less than 12 g/dL
* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) value greater than twice the upper limit of the normal range (ULN)
* total bilirubin value of more than 25.7 μmol/L (1.5 mg/dL)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Drug Liking and Effects Questionnaire (DLEQ) | Phase B: prior to and at designated times up to 24 hours after study drug administration. Phase C:prior to and at set times up to 72 hours after study drug administration
  The DLEQ measures positive, negative, and any drug effects using bipolar and unipolar VAS. Bipolar VAS range from a strong negative response (score of 0) to a strong positive response (score of 100) with a neutral midpoint (score of 50). Unipolar VAS range from a response of 'none' (score of 0) to 'extremely' (score of 100). Questions include assessments of liking, drowsiness, good effects, bad effects, nausea,and any effects. The primary outcome is question 1 which states: "My liking for this drug is:"

SECONDARY OUTCOMES:
Overall drug liking visual analog scale (VAS) score | 24 hours after the start of each study drug administration in phase B and C
  Overall drug liking scale measures the extent the subject "likes" the drug as measured on a 100 mm visual analog scale anchored at one end by the phrase "strong disliking" and on the other end by "strong liking", and in the middle (50 mm) "neither like nor dislike". The question posed to the subject is: "overall, my liking for this drug is:".
Pharmacokinetic maximum observed (Cmax) plasma concentrations | Approximately 30 minutes before study drug administration up to 72 hours post study drug administration
  To characterize the pharmacokinetics of the hydrocodone bitartrate extended-release tablet (crushed and intact) and immediate-release hydrocodone bitartrate by assessing plasma concentration data over 72 hours following study drug administration
Take drug again Visual Analog Scale | 24 hours after the start of each study drug administration in phase B and C
  Take drug again visual analog scale measures the extent the subject is willing to take the drug again as measured on a 100 mm visual analog scale anchored at one end by the phrase "Definitely would not" and on the other end by "definitely would". The question posed to the subject is: "If given the opportunity, I would want to take this drug again:".
Price Value Assessment Questionnaire | 24 hours after the start of each study drug administration in phase B and C
  Price Value Assessment Questionnaire measures the subjective assessment of perceived value of a drug. The question posed to the subject is: "What is the most that you would be willing to pay for the same dose of the drug that you have just taken, if it was offered to you on the street?" The subject chooses from a list of dollar amounts. The greater the dollar amount the more the subject values the drug.
Addiction Research Center Inventory (ARCI): Morphine Benzedrine Group (MBG) Subscale | Phase B: prior to and at designated times up to 24 hours after study drug administration. Phase C:prior to and at set times up to 72 hours after study drug administration
  The Addiction Research Center Inventory (ARCI) is a questionnaire consisting of several distinct subscales that assesses mood states typically associated with certain classes of drugs through the use of true or false questions. The Morphine Benzedrine Group (MBG) subscale assesses euphoria with 16 true or false questions. Each true item is given a score of 3 and each false item is scored 0. Higher scores are associated with greater euphoria. Minimum score is 0, highest score is 48.
Addiction Research Center Inventory (ARCI): Lysergic Acid Diethylamide (LSD) Subscale | Phase B: prior to and at designated times up to 24 hours after study drug administration. Phase C:prior to and at set times up to 72 hours after study drug administration
  The Addiction Research Center Inventory (ARCI) is a questionnaire consisting of several distinct subscales that assesses mood states typically associated with certain classes of drugs through the use of true or false questions. The Lysergic Acid Diethylamide (LSD) subscale assesses dysphoria with 14 true or false questions. Each true item is given a score of 3 and each false item is scored 0. Higher scores are associated with greater dysphoria. Minimum score is 0, highest score is 42.
Addiction Research Center Inventory (ARCI): Pentobarbital Chlorpromazine Alcohol Group (PCAG) Subscale | Phase B: prior to and at designated times up to 24 hours after study drug administration. Phase C:prior to and at set times up to 72 hours after study drug administration
  The Addiction Research Center Inventory (ARCI) is a questionnaire consisting of several distinct subscales that assesses mood states typically associated with certain classes of drugs through the use of true or false questions. The Pentobarbital Chlorpromazine Alcohol Group (PCAG) Subscale assesses sedation with 15 true or false questions. Each true item is given a score of 3 and each false item is scored 0. Higher scores are associated with greater dysphoria. Minimum score is 0, highest score is 45.
Pupillometry | Phase B: prior to and at designated times up to 24 hours after study drug administration. Phase C:prior to and at set times up to 72 hours after study drug administration
  Pupillometry measures change in pupil size (miosis - shrinkage of pupil) as an indicator of opioid pharmacological properties. The same eye for each subject will be used for all measurements during the study.
Time to maximum observed drug concentration (tmax) | Approximately 30 minutes before study drug administration up to 72 hours post study drug administration
  To characterize the pharmacokinetics of the hydrocodone bitartrate extended-release tablet (crushed and intact) and immediate-release hydrocodone bitartrate by assessing plasma concentration data over 72 hours following study drug administration
Area under the plasma concentration by time curve (AUC) from time 0 to maximum drug concentration time - Immediate release product | Approximately 30 minutes before study drug administration up to 72 hours post study drug administration
  To characterize the pharmacokinetics of the hydrocodone bitartrate extended-release tablet (crushed and intact) and immediate-release hydrocodone bitartrate by assessing plasma concentration data over 72 hours following study drug administration
Area under the plasma concentration by time curve (AUC) from time 0 to maximum drug concentration time - Extended release product intact | Approximately 30 minutes before study drug administration up to 72 hours post study drug administration
  To characterize the pharmacokinetics of the hydrocodone bitartrate extended-release tablet (crushed and intact) and immediate-release hydrocodone bitartrate by assessing plasma concentration data over 72 hours following study drug administration
Area under the plasma concentration by time curve (AUC) from time 0 to maximum drug concentration time - Extended release product crushed | Approximately 30 minutes before study drug administration up to 72 hours post study drug administration
  To characterize the pharmacokinetics of the hydrocodone bitartrate extended-release tablet (crushed and intact) and immediate-release hydrocodone bitartrate by assessing plasma concentration data over 72 hours following study drug administration
Area under the plasma concentration by time curve (AUC) from time 0 to last measureable drug concentration | Approximately 30 minutes before study drug administration up to 72 hours post study drug administration
  To characterize the pharmacokinetics of the hydrocodone bitartrate extended-release tablet (crushed and intact) and immediate-release hydrocodone bitartrate by assessing plasma concentration data over 72 hours following study drug administration
Area under the plasma concentration by time curve (AUC) from time 0 to infinity | Approximately 30 minutes before study drug administration up to 72 hours post study drug administration
  To characterize the pharmacokinetics of the hydrocodone bitartrate extended-release tablet (crushed and intact) and immediate-release hydrocodone bitartrate by assessing plasma concentration data over 72 hours following study drug administration
Apparent plasma terminal elimination rate constant and associated elimination half-life | Approximately 30 minutes before study drug administration up to 72 hours post study drug administration
  To characterize the pharmacokinetics of the hydrocodone bitartrate extended-release tablet (crushed and intact) and immediate-release hydrocodone bitartrate by assessing plasma concentration data over 72 hours following study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Cephalon
Locations (2):
- Cephalon Investigational Site 001, Salt Lake City, Utah, United States
- Cephalon Investigational Site 100, Toronto, Ontario, Canada